CLINICAL TRIAL: NCT01478776
Title: The Impact of Omega-3 Supplementation on Acylation Stimulating Protein(ASP), Retinol-binding Protein 4 (RBP4) and Lipocalin-2 (LCN2) Gene Expression of ASP Receptor (C5L2) in WBC of Patient With Diabetes Type 2
Brief Title: The Impact of Omega-3 Supplementation on Gene Expression in Type 2 Diabetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15176
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes
Keywords: ASP; LCN2; RBP4; C5L2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- diabetes, omega-3 (Active Comparator): patient with type 2 diabetes who receive 4gr/day omega-3
  Interventions: Dietary Supplement: omega-3
- placebo, diabetes (Placebo Comparator): patient with type 2 diabetes who receive 4 cap of placebo/day
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 — 4 cap 1 gr omega-3 per day for 10 weeks
  Other Names: n-3 fatty acids,n-3 PUFA
  Arms: diabetes, omega-3
Dietary Supplement: placebo — patient with type 2 diabetes who receive 4 cap placebo/day for 10 weeks
  Arms: placebo, diabetes

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with omega-3 or placebo for 10 weeks in type 2 diabetics

DETAILED DESCRIPTION:
Adipose tissue is recognized as an important endocrine organ in human. Not only it has function of storing unlimited energy but also its secretory roles is subject to intense research in recent years. Acylation stimulating protein(ASP), Retinol-binding protein 4 (RBP4) and lipocalin-2 (LCN2) are circulating adipokines elevated in diabetes. C5L2 is a G-protein-coupled receptor. activation of C5L2 by ASP, has been shown. Fatty acids may influence the expression of adipokines. Epidemiological studies showed that omega-3 reduce the development of insulin resistance and diabetes. Because fatty acids are the main component of adipose tissue, it is essential interest to clarify the biological effects of omega-3 on the expression of relevant adipokines.

ELIGIBILITY:
Inclusion Criteria:

* literate
* Willingness to participation
* Diabetic patients 30-65 years old
* Body mass index in the range 18.5-40
* Avoidance of dietary supplements
* vitamins and herbal products at least 2 weeks before and throughout the intervention

Exclusion Criteria:

* people who have used omega-3 supplements in last 3 months
* Having chronic renal disease
* hepatic disease
* gastrointestinal disease
* hematological disorders
* hypothyroidism or hyperthyroidism
* Treatment with Orlistat or sibutramine for weight loss
* Pregnancy and lactation
* Treatment with insulin or Thiazolidinediones

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
serum total cholesterol | change from baseline at 10 weeks
serum High-density lipoprotein (HDL) cholesterol | change from baseline at 10 weeks
serum Low-density lipoprotein (LDL) cholesterol | change from baseline at 10 weeks
serum triglycerides (TG) level | change from baseline at 10 weeks
postprandial triglycerides | change from baseline at 10 weeks
complete blood count(CBC) | change from baseline at 10 weeks
fasting plasma glucose(FPG) | change from baseline at 10 weeks
Glycated hemoglobin (Hb A1c) | change from baseline at 10 weeks
acylation stimulating protein (ASP) | change from baseline at 10 weeks
lipocalin-2 (LCN2) | change from baseline at 10 weeks
Retinol-binding protein 4 (RBP4) | change from baseline at 10 weeks
non-esterified fatty acids (NEFA) | change from baseline at 10 weeks
insulin | change from baseline at 10 weeks
postprandial ASP | chage from baseline at 10 weeks

SECONDARY OUTCOMES:
gene expression of C5L2 | change from baseline at 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Tehran Province, Iran